CLINICAL TRIAL: NCT06352047
Title: The Effects of Positioning After Extubation of Preterm Infants on the Respiratory Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, İlknur KAHRİMAN, Associate Prof. Dr, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Karadeniz Tech. University
Record Dates: First submitted 2024-03-17; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Premature Infants
Keywords: Extubation; Position; Premature; Supine; Prone
MeSH Terms: conditions — Premature Birth; Deception

STUDY DESIGN:
Intervention Model Description: Simple randomization method was used in the sample of the study. In previous studies, there were no published data on the effect of supine and prone positioning after extubation on the pulmonary functions of premature infants. Therefore, the sample size was calculated using the G-power 3.1.3 program according to the SpO2 level and standard deviation values of 4 infants who were mechanically ventilated in the neonatal intensive care unit. The study was conducted with a total of 42 premature babies, two groups of 21 premature babies, each of whom had the characteristics of the research groups. Premature infants were divided into two groups, the supine position and the prone group, by randomization using a computer-based random number generator (www.randomizer.org).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine position group (Experimental): Supine position group Before starting the study, parents of preterm infants were informed about the study, and the infants of parents who agreed to participate in the study were divided into two groups as prone and supine positions. In the study, preterm babies positioned after extubation by the researcher. Before extubation, SpO2, respiratory rate (to be counted for one minute), blood pressure, blood gas values were checked and recorded from the bedside monitor of the babies planned for extubation. Before leaving the mechanical ventilator for preterm newborns who were decided for extubation and met the research criteria, vibration and percussion were performed to premature babies over 1500 g with a mouth mask or palm dome. Oral, nasal and oranazopharynx were aspirated for 3-5 seconds with an appropriate aspiration catheter (6-8 Fr) at a pressure not exceeding 100 mmHg.
  Interventions: Other: The effect of positioning on respiratory functions of preterm infants after extubation.
- Prone position group (Active Comparator): Prone position group Before starting the study, parents of preterm infants were informed about the study, and the infants of parents who agreed to participate in the study were divided into two groups as prone and supine positions. In the study, preterm babies positioned after extubation by the researcher. Before extubation, SpO2, respiratory rate (to be counted for one minute), blood pressure, blood gas values obtained from the heel blood of the Preterm baby were checked on the bedside monitor and recorded before extubation. Before leaving the mechanical ventilator for preterm newborns who were decided for extubation and met the research criteria, vibration and percussion were performed to premature babies over 1500 g with a mouth mask or palm dome. Oral, nasal and oranazopharynx were aspirated for 3-5 seconds with an appropriate aspiration catheter (6-8 Fr) at a pressure not exceeding 100 mmHg.
  Interventions: Other: The effect of positioning on respiratory functions of preterm infants after extubation.

INTERVENTIONS:
Other: The effect of positioning on respiratory functions of preterm infants after extubation. — Position changes and the direction of the position (supine, prone, side lying) are recorded in the nurse observation form.

SUMMARY:
The aim of this study was to examine the effect of positioning on respiratory functions of preterm infants after extubation.

Hypothesis 0a (H0a): There is no difference between the oxygen saturation (SpO2) levels of preterm infants in supine and prone positions after extubation.

Hypothesis 0b (H0b): There is no difference between the respiratory rate of preterm infants in supine and prone positions after extubation.

Hypothesis 0c (H0c): There is no difference between the respiratory rhythms of preterm infants in supine and prone positions after extubation.

Hypothesis 0d (H0d): There is no difference between respiratory distress in preterm infants in supine and prone positions after extubation.

DETAILED DESCRIPTION:
Among infants in the neonatal intensive care unit (NICU), the ones in the high and medium risk group are premature infants. Respiratory distress is the most important problem in infants with a history of preterm birth due to undeveloped systems and organs. Especially premature infants need respiratory support in the NICU. The most important stage of supportive treatment is the application of mechanical ventilation with endotracheal intubation. Newborns receiving mechanical ventilation support should be checked constantly Considering that endotracheal intubation may cause extreme stress and traumatic effects on premature babies, it should be ensured that premature babies get through the ventilation process and afterward with minimal trauma. This will positively affect the adaptation process after the termination of intubation. The neonatal nurse continuously monitors the changes in heart rate, body temperature, blood pressure, SpO2, respiratory characteristics and number of infants receiving mechanical ventilation and records them in the patient follow-up form. The nurse tries to provide the most ideal respiratory form in infants with mechanical ventilation. For this reason, neonatal nurses should provide individualized developmental nursing care by considering all the physiological needs of premature babies in order to provide the most ideal respiratory form. The use of individualized care models in premature babies increases the health quality and social cohesion of preterm babies. It fastens the physiological recovery, shortens the hospital stay and increases neurodevelopmental functions. Positionig is one of the most important developmental supportive activities. It is important in nursing care to position the preterm babies appropriately and to ensure its continuity according to their needs. It is recommended that preterm infants with respiratory distress in the NICU should be placed in the supine position after extubation when respiratory patterns are stabilized. It has been observed that the prone position increases oxygen saturation in premature babies, shortens the duration of mechanical ventilator therapy, decreases re-intubation after extubation, decreases neonatal apnea, and contributes to the development of respiratory muscles and positively affects respiratory functions. In addition, the prone position increases the lung capacity of preterm infants. Studies show that the prone position improves diaphragmatic function, increases lung perfusion, and has positive effects on respiratory functions. In another study, it was stated that the prone position is a safe and healthy process according to the order of separation from mechanical ventilation and may contribute to the success of separation from mechanical ventilation in preterm infants [4]. The neonatal nurse should be aware of the importance of positioning and should be able to position the newborn baby when needed in routine care practices. During the respiratory system intubation period and after extubation, the effects of the positioning on the respiratory functions of the preterm should be observed and the position with the highest benefit should be taken into consideration when performing individualized nursing care. Therefore, the aim of this study was to examine the effect of positioning on respiratory functions of preterm infants after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheal intubation was applied,

  * Those whose gestational weeks are under 37+6 years of age,
  * Parts of premature babies whose parents gave written consent to participate were included.

Exclusion Criteria:

* Developing pneumothorax,

  * Those with congenital anomalies,
  * Those with intracranial hemorrhage and/or periventricular leukomalacia,
  * Surgery that may affect heart, circulation and respiratory functions or prevent supine/prone positioning,
  * Not intubated,
  * Premature babies whose parents gave up participating in the study were not included in the study.

Ages: 37 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Newborn Evaluation Form | 120 minutes
  After the positioning, vital measurements (fever, HR, blood pressure), respiratory characteristics (number, rhythm, distress), SpO2 values were recorded. These infants were monitored for 120 minutes. Every 30 minutes, respiratory rate, HR, SpO2 were evaluated from the bedside monitor. After 60 minutes, blood gas parameters were evaluated. The presence of desaturation, apnea, and cyanosis was observed within 120 minutes and recorded in the data collection forum. During this process, the researcher stayed with the baby and recorded the measurement results and other observed findings on the observation form.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İlknur Kahriman, Trabzon
  - Karadeniz Technical University Health Application and Research Center Farabi Hospital, Trabzon

IPD SHARING:
Plan to Share IPD: No